CLINICAL TRIAL: NCT06683417
Title: Vestibular Rehabilitation Aid (VestAid)
Brief Title: Effectiveness of VestAid App
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BlueHalo (Industry)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24060038
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: MTBI - Mild Traumatic Brain Injury; Vestibular Disease; Balance Deficits; Vestibular Disorders; Dizziness
Keywords: mTBI; vestibular rehabilitation; vestibular disorder; technology; application; dizziness; balance disorder; image processing; eye gaze compliance; VOR
MeSH Terms: conditions — Brain Concussion; Vestibular Diseases; Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- VestAid (Experimental): Use of VestAid tablet application to aid vestibular rehabilitation
  Interventions: Device: Vestibular Rehabilitation Aid
- Standard of Care vestibular rehabilitation (Active Comparator): Use of standard of care vestibular rehabilitation
  Interventions: Other: Standard of care vestibular rehabilitation

INTERVENTIONS:
Device: Vestibular Rehabilitation Aid — The tablet-based VestAid system was developed to repair, restore and maintain vestibular-ocular function that is impaired in patients post-mTBI.
  Each participant's treating physical therapist will develop their own personalized exercise prescription. The physical therapist will be asked to recommend that the patients complete a home exercise program at least 2-3 times per day for 6 weeks. The exercise prescription will be placed on the VestAid by the physical therapist for the patient to follow. The patient is not able to modify the exercise, only the physical therapist can modify the exercises. Exercises will be modified based on patient's response and symptom reports. The physical therapist and study coordinator will receive an alert on the VestAid online dashboard if the patient's symptoms are greater than or equal to 8/10.
  Other Names: VestAid
  Arms: VestAid
Other: Standard of care vestibular rehabilitation — Vestibular rehabilitation to include gaze stabilization exercises, optokinetic training, smooth pursuits and saccades
  Arms: Standard of Care vestibular rehabilitation

SUMMARY:
This multi-center randomized trial (MCRT) will investigate the effectiveness of the VestAid application to provide equivalent or faster recovery from dizziness compared to standard-of-care delivery of vestibular rehabilitation exercises.

ELIGIBILITY:
Inclusion:

* Snellen visual acuity (corrected) greater than 20/40
* No more than 25dB hearing loss at 500,1000, 2000, and 4000 Hz
* Ability to detect 4.31 using Semmes-Weinstein monofilament at the lower extremity
* At least 40 degrees of neck yaw motion with only mild to moderate pain (6 or under on 0-10 numeric pain scale)
* Internet access at home
* No significant residual from past musculoskeletal or neuromuscular conditions
* Ability ambulates unassisted
* Diagnosed with a concussion or inner ear problem the last 30 days
* Between 18-60 years of age
* Can read and understand English
* Has complaints of dizziness

Exclusion criteria:

* Greater then 30 days since diagnosis of concussion/mTBI or inner ear problem
* No access to internet at home
* Younger than 18 years of age or older than 60 years of age
* Cannot read or understand English
* No complaints of dizziness and/or balance deficits
* Have significant neuropathy
* Cannot see tablet clearly at 1 meter
* Neck pain >5 on a 10-point pain scale.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | From enrollment weekly for 6 weeks.
  A self report measure of dizziness (questionnaire)

SECONDARY OUTCOMES:
Secondary Endpoint | From enrollment weekly for 6 weeks
  Subjective symptom reporting of dizziness, headache, nausea, and fogginess

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Whitney SL, Sparto PJ. Principles of vestibular physical therapy rehabilitation. NeuroRehabilitation. 2011;29(2):157-66. doi: 10.3233/NRE-2011-0690. PMID 22027077
- [Background] Shepard NT, Telian SA. Programmatic vestibular rehabilitation. Otolaryngol Head Neck Surg. 1995 Jan;112(1):173-82. doi: 10.1016/S0194-59989570317-9. PMID 7816453
- [Background] Gottshall K. Vestibular rehabilitation after mild traumatic brain injury with vestibular pathology. NeuroRehabilitation. 2011;29(2):167-71. doi: 10.3233/NRE-2011-0691. PMID 22027078
- [Background] Hall CD, Herdman SJ. Reliability of clinical measures used to assess patients with peripheral vestibular disorders. J Neurol Phys Ther. 2006 Jun;30(2):74-81. doi: 10.1097/01.npt.0000282571.55673.ed. PMID 16796772
- [Background] Essery R, Geraghty AW, Kirby S, Yardley L. Predictors of adherence to home-based physical therapies: a systematic review. Disabil Rehabil. 2017 Mar;39(6):519-534. doi: 10.3109/09638288.2016.1153160. Epub 2016 Apr 21. PMID 27097761
- [Background] Mucha A, Collins MW, Elbin RJ, Furman JM, Troutman-Enseki C, DeWolf RM, Marchetti G, Kontos AP. A Brief Vestibular/Ocular Motor Screening (VOMS) assessment to evaluate concussions: preliminary findings. Am J Sports Med. 2014 Oct;42(10):2479-86. doi: 10.1177/0363546514543775. Epub 2014 Aug 8. PMID 25106780